CLINICAL TRIAL: NCT01553305
Title: The Effect of 6-weeks Supervised Exercise Programme Followed by 6-weeks Unsupervised Exercise Programme Versus 12 Weeks Unsupervised Exercise Programme in Patients With Rheumatoid Arthritis.
Brief Title: A Study of the Effect of Supervised Exercise Programme in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Trine Seneca, Physiotherapist, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AarhusUH-TS; AarhusUH-TS
Record Dates: First submitted 2012-03-04; First posted 2012-03-14 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: exercise programme
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised exercise programme (Experimental): Six-weeks supervised high-intensity exercise programme with training sessions twice a week followed by 6-weeks unsupervised exercise programme.
  Interventions: Other: Supervised high-intensity exercise programme; Other: Exercise programme
- Unsupervised exercise programme (No Intervention)

INTERVENTIONS:
Other: Supervised high-intensity exercise programme — Six-weeks supervised high-intensity muscle strength training and physical fitness with training sessions twice a week followed by 6-weeks unsupervised high-intensity exercise programme.
  Arms: Supervised exercise programme
Other: Exercise programme — Supervised exercise programme
  Arms: Supervised exercise programme

SUMMARY:
The purpose of this study is to compare the effectiveness of a supervised high-intensity exercise programme followed by an unsupervised exercise programme to an unsupervised exercise programme in patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Patients with Rheumatoid Arthritis are in general less fit and more at risk of comorbidities such as cardiovascular events compared with healthy age-matched controls. Studies indicates that patients with Rheumatoid Arthritis have a lower level of physical activity than the general population and a low proportion of patients with Rheumatoid Arthritis exercises. Regular exercise with moderate to high intensity level of intensity has proven to be effective in reducing the cardiovascular risk by improving cardiovascular fitness and to increase muscle strength. Therefore, it is of interest to investigate if supervised exercise programme makes a difference making patients with Rheumatoid Arthritis participate in exercise.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Rheumatoid Arthritis within the last three years at Aarhus University Hospital according to the 1987 revised ACR criteria or the 2009 ACR/EULAR criteria
* must be able to sit on an exercise bike
* must be able to participate in 6-weeks exercise programme with training sessions twice a week at Aarhus University Hospital
* must be able to speak and understand danish

Exclusion Criteria:

* high disease activity assessed by DAS28-CRP
* Myocardial Infarction within the last six months
* Angina Pectoris
* treated with beta-blocker
* severe high blood pressure
* severe lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength (kg) | Muscle strength is measured at baseline and follow-up. The outcome is change in muscle strength in 12 weeks from baseline to follow-up.

SECONDARY OUTCOMES:
Change in cardiovascular fitness | Cardiovascular fitness is measured at baseline and follow-up. The outcome is change in cardiovascular fitness in 12 weeks from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Seneca, Principal Investigator — Aarhus University Hospital, Department of Physiotherapy
Locations (1):
- Aarhus University Hospital, Department of Physiotherapy, Aarhus, Denmark

REFERENCES:
- [Derived] Seneca T, Hauge EM, Maribo T. Comparable effect of partly supervised and self-administered exercise programme in early rheumatoid arthritis--a randomised, controlled trial. Dan Med J. 2015 Aug;62(8):A5127. PMID 26239594